CLINICAL TRIAL: NCT03041792
Title: A 6-WEEK, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, TWO-ARM, PARALLEL METHODOLOGY STUDY TO ASSESS THE EFFECT OF LIRAGLUTIDE ON FOOD INTAKE IN OBESE SUBJECTS
Brief Title: Methodology Study To Examine 6-Week Food Intake With Liraglutide In Obese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: A9001498
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Liraglutide
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Liraglutide — Liraglutide
  Arms: Active
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This will be a randomized, double blind, placebo controlled, 2 arm, parallel group, methodology study to assess the effect of 6 weeks of liraglutide administration on food intake in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males and female subjects;
* Body Mass Index 30-40 kg/m2;

Exclusion Criteria:

* Evidence of history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergises, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001498&StudyName=A+6-WEEK%2C+RANDOMIZED%2C+DOUBLE-BLIND%2C+PLACEBO-CONTROLLED%2C+TWO-ARM%2C+PARALLEL+METHODOLOGY+STUDY+TO+ASSESS+THE+EFFECT+OF+LIRAGLUTIDE+ON+FOOD+INTAKE+IN+OBESE+SUBJECTS

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, a total of 61 potential participants were randomized to the study, and 60 of them received study treatment.
Groups:
- Liraglutide: Liraglutide was administered subcutaneously via pen injection with dose titration to 3.0 milligram (mg) daily per Saxenda prescribing instructions.
- Placebo: 0.9% weight/volume (w/v) sodium chloride, United States Pharmacopeia (USP), was administered subcutaneously as placebo via syringe injection daily with matching volume to liraglutide dose.
Period: Overall Study
Arm/Group | Liraglutide | Placebo
Started | 32 | 29
Received Treatment | 32 | 28
Completed | 28 | 26
Not Completed | 4 | 3
Not completed — Adverse Event | 4 | 0
Not completed — Death in the family | 0 | 2
Not completed — Randomized but not treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who met the criteria stated below were included in the full analysis set (FAS): completed baseline assessment of food intake; received at least one dose of randomized, blinded investigational product (IP); and completed at least one post baseline measurement (after taking randomized IP).
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide | Placebo | Total
Number analyzed (Participants) | 30 | 26 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (10.88) | 48.1 (12.63) | 45.4 (11.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 16 | 38
  Male | 8 | 10 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21 | 19 | 40
  Black or African American | 9 | 6 | 15
  Asian | 0 | 1 | 1
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 0 | 0 | 0
  Unknown | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Visit 3) in Mean Energy Intake During Ad Libitum Lunches at Visits 4 and 5
Description: The mean energy intake was collected to assess the effect of liraglutide on food intake in non-diabetic, obese participants. Observed food intake was measured as the total number of calories consumed during the specified time period, calculated as the difference of the total number of calories provided minus the total number of calories remaining after meals. Mean energy intakes at Visit 4 was defined as the mean values of the measurements at Study Day 20 and 21. Same definition applies to Visit 5 (Study Day 41 and 42). Baseline was defined as the mean of Visit 3 (Study Day -1 and 0).
Time Frame: Visit 3, Visit 4 and Visit 5
Population: Number of participants analyzed includes participants who met the criteria: completed baseline assessment of food intake;received at least 1 dose of randomized, blinded IP;completed at least 1 post baseline measurement(after taking randomized IP).Number analyzed includes participants contributing to mean energy intake at specified visits.
Measure: Mean (Standard Deviation); unit: kilocalories (kcal)
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 30 | 26
kilocalories (kcal)
  Visit 4 | -254.48 (160.67) | -19.93 (162.12)
  Visit 5: number analyzed (Participants) | 28 | 26
  Visit 5 | -278.78 (190.09) | -37.43 (164.49)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Visit 4; Test type: Superiority; p = 0.0000, Mixed Models Analysis — The p-value was calculated and was rounded to 4th decimal presenting as 0.0000, which was smaller than the required threshold of <0.05; Least Square Mean Difference = -235.75, 95% CI 2-sided [-322.25 to -149.25], Standard Error of Mean 43.13
Statistical Analysis 2: Comparison: Liraglutide vs Placebo; Visit 5; Test type: Superiority; p = 0.0000, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Least Square Mean Difference = -243.63, 95% CI 2-sided [-339.10 to -148.15], Standard Error of Mean 47.60

2. Secondary Outcome: Number of Participants With Vital Signs Data Meeting Categorical Criteria
Description: Absolute values and changes from baseline in systolic blood pressure (SBP) and diastolic blood pressure (DBP), pulse rate (PR) were recorded in supine position. Vital signs categorical summarization criteria were 1), blood pressure: SBP greater than or equal to (>=) 30 millimeters of mercury (mm Hg) change from baseline, SBP less than (<) 90 mm Hg; DBP >=20 mm Hg change from baseline, DBP <50 mm Hg; 2), PR <40 or greater than (>) 120 beats per minute (bpm). Baseline was defined as pre-treatment measurement on Day 1.
Time Frame: Baseline (Visit 3) up to Visit 6 (Study Day 53)
Population: All participants who received at least 1 dose of study medication classified according to the actual study treatment received. Follow-up readings have been excluded from presentation, and 4 participants have been excluded from presentation because they only have follow up readings in post-dose phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 30 | 26
Participants
  Supine DBP <50 mmHg | 3 | 5
  Supine PR <40 bpm | 0 | 0
  Supine PR >120 bpm | 0 | 0
  Supine SBP <90 mmHg | 1 | 2
  Increase in supine DBP >=20 mmHg | 3 | 1
  Increase in supine SBP >=30 mmHg | 1 | 1
  Decrease in supine DBP >=20 mmHg | 3 | 9
  Decrease in supine SBP >=30 mmHg | 1 | 0

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (All-Causality)
Description: Adverse event (AE) was defined as any untoward medical occurrence in a study participant administered a product or medical device, regardless of its causal relationship with study treatment. An AE is considered treatment-emergent relative to a given treatment if: the event occurs for the first time during the effective duration of treatment and was not seen prior to the start of treatment (for example, during the baseline or run-in period); or the event was seen prior to the start of treatment but increased in severity during treatment.
Time Frame: Baseline (Visit 3) up to 31 days post last dose (75 days)
Population: The safety analysis population included all participants who received at least one dose of study medication classified according to the actual study treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 31 | 20

4. Secondary Outcome: Number of Participants With Abnormal 12-lead Electrocardiogram (ECG)
Description: ECG categorical summarization criteria: 1) PR interval (the interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization): absolute value greater than or equal to (>=) 300 msec, percent change >=25% if baseline was greater than (>) 200 msec, and >=50% if baseline was less than or equal to (<=) 200 msec; 2) QRS interval (time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization): absolute value >=200 msec, percent change >=25% if baseline was 100 msec, and >=50% if baseline was <=100 msec; 3) QTcF interval (QT corrected for heart rate using Fridericia's formula): absolute value >450 to <=480 msec, >480 to <=500 msec, >500 msec, an increase from baseline >30 to <=60 msec or >60 msec. Baseline was defined as pre-treatment measurement on Day -2.
Time Frame: Baseline (Visit 3) up to Visit 6 (Study Day 53)
Population: All participants who received at least one dose of study medication classified according to the actual study treatment received. Follow-up readings have been excluded from presentation, and 4 participants have been excluded from presentation because they only have follow up readings in post-dose phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 30 | 26
Participants
  PR interval >=300 milliseconds (msec) | 0 | 0
  QRS interval >=200 msec | 0 | 0
  QTcF >450 - <=480 msec | 2 | 2
  QTcF >480 - <=500 msec | 0 | 0
  QTcF >500 msec | 0 | 0
  PR interval percent increase >=25/50% | 0 | 0
  QRS interval percent increase >=25/50% | 0 | 0
  QTcF increase >30 - <=60 msec | 2 | 1
  QTcF increase >60 msec | 0 | 0

5. Secondary Outcome: Number of Participants With Laboratory Abnormalities (Without Regard to Baseline Abnormality)
Description: Below parameters were evaluated:1), Hematology: hemoglobin (HGB), hematocrit, erythrocytes (absolute value/mean corpuscular volume/mean corpuscular HGB/mean corpuscular HGB concentration), platelets, leukocytes, lymphocytes, neutrophils, basophils, monocytes; 2), clinical chemistry: bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, protein, albumin, blood urea nitrogen, creatinine, cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, triglycerides, sodium, potassium, chloride, calcium, bicarbonate, amylase, triacylglycerol lipase; 3), urinalysis: pH, urine glucose, ketones, urine protein, urine hemoglobin, urobilinogen, urine bilirubin, nitrite, leukocyte esterase, urine erythrocytes, urine leukocytes, hyaline casts, bacteria.
Time Frame: Baseline (Visit 3) up to Visit 6 (Study Day 53)
Population: All participants who received at least one dose of study medication classified according to the actual study treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 32 | 28
Participants | 32 | 26

6. Secondary Outcome: Change From Baseline in Mean 48-hour Energy Intake at Visits 4 and 5
Description: Energy intake was measured over a period of 48 hours to assess day to day variability in food intake. Observed food intake was measured as the total number of calories consumed during the specified time period, calculated as the difference of the total number of calories provided minus the total number of calories remaining after meals. Baseline was defined as the 48 hour period at Visit 3 (Study Day -1 and 0).
Time Frame: Visit 3, Visit 4 (Study Day 20 and 21) and Visit 5 (Study Day 41 and 42)
Population: Number of participants analyzed includes participants who met the criteria: completed baseline assessment of food intake;received at least 1 dose of randomized, blinded IP;completed at least 1 post baseline measurement(after taking randomized IP).Number analyzed includes participants contributing to mean 48-hour energy intake at specified visits.
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 30 | 26
kcal
  Visit 4 | -1058.8 (627.61) | -205.64 (608.51)
  Visit 5: number analyzed (Participants) | 28 | 26
  Visit 5 | -1152.5 (745.71) | -242.84 (681.37)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Visit 4; Test type: Superiority; p = 0.0000, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Least Square Mean Difference = -859.58, 95% CI 2-sided [-1196.1 to -523.10], Standard Error of Mean 167.76
Statistical Analysis 2: Comparison: Liraglutide vs Placebo; Visit 5; Test type: Superiority; p = 0.0000, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Least Square Mean Difference = -928.56, 95% CI 2-sided [-1317.3 to -539.86], Standard Error of Mean 193.80

7. Secondary Outcome: Change From Baseline in Appetite Score (Mean Rating Area Under Curve From Time 30 to 120 Minutes [AUC30-120min]) for Mean Lunch at Visits 4 and 5
Description: Appetite, satiety, fullness, hunger, and prospective consumption were measured using a validated Visual Analog scale (VAS) questionnaire. VAS was an assessment in which participants place a vertical line across a validated 100 millimeter (mm) line with the example of "Not At All Full" and "Totally Full" at either end, scoring from 0 to 100. The overall appetite score was calculated as the average of the four individual scores [satiety + fullness + (100 - prospective food consumption)+(100 - hunger)] divided by 4. The VAS questionnaire was completed by the participant immediately prior to meal administration, and at 30, 60 and 120 minutes after start of the specified meals. Baseline of Mean Rating AUC30-120min was defined as the rating for mean lunch at Visit 3 (Study Day -1 and 0).
Time Frame: Visit 3, Visit 4 (Study Day 20 and 21) and Visit 5 (Study Day 41 and 42)
Population: Number of participants analyzed includes participants who met the criteria: completed baseline assessment of food intake;received at least 1 dose of randomized, blinded IP;completed at least 1 post baseline measurement(after taking randomized IP).Number analyzed includes participants contributing to appetite score at specified visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 30 | 26
units on a scale
  Visit 4: number analyzed (Participants) | 28 | 26
  Visit 4 | 4.52 (8.65) | -0.60 (9.22)
  Visit 5: number analyzed (Participants) | 28 | 26
  Visit 5 | 4.13 (9.99) | -0.99 (8.17)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Visit 4; Test type: Superiority; p = 0.0263, Mixed Models Analysis; Least Square Mean Difference = 4.95, 95% CI 2-sided [0.61 to 9.29], Standard Error of Mean 2.16
Statistical Analysis 2: Comparison: Liraglutide vs Placebo; Visit 5; Test type: Superiority; p = 0.0121, Mixed Models Analysis; Least Square Mean Difference = 5.35, 95% CI 2-sided [1.22 to 9.48], Standard Error of Mean 2.06

8. Secondary Outcome: Change From Baseline in Satiety, Fullness, Prospective Food Consumption and Hunger Scores (Mean Rating AUC30-120min) for Mean Lunch at Visits 4 and 5
Description: Satiety, fullness, hunger, and prospective consumption were measured at the study site using a validated VAS questionnaire. The VAS measurement of the subcomponent scores were the same as that of the appetite score. Baseline of Mean Rating AUC30-120min was defined as the rating for mean lunch at Visit 3 (Study Day -1 and 0).The VAS was an assessment in which subjects place a vertical line across a validated 100 millimeter (mm) line to rank their response to various questions. The line was anchored by responses such as "Not At All Full" and "Totally Full" at either end. Scoring consisted of measuring the distance in mm of the vertical line from the response at the left end. The scores (total and subscale) ranged from 0 to 100. The lower values represent the better outcomes.The overall appetite score was calculated as the average of the 4 individual scores [satiety+fullness+(100-prospective food consumption)+(100-hunger)] divided by 4.
Time Frame: Visit 3, Visit 4 (Study Day 20 and 21) and Visit 5 (Study Day 41 and 42)
Population: Number of participants analyzed includes participants who met the criteria: completed baseline assessment of food intake;received at least 1 dose of randomized, blinded IP;completed at least 1 post baseline measurement(after taking randomized IP).Number analyzed includes participants contributing to VAS scores at specified visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 30 | 26
units on a scale
  Satiety (Visit 4) | 3.94 (13.50) | -0.55 (10.52)
  Satiety (Visit 5): number analyzed (Participants) | 28 | 26
  Satiety (Visit 5) | 4.51 (11.79) | 1.02 (9.26)
  Fullness (Visit 4) | 4.04 (9.52) | 1.88 (10.85)
  Fullness (Visit 5): number analyzed (Participants) | 28 | 26
  Fullness (Visit 5) | 2.40 (10.08) | 1.89 (9.17)
  Prospective food consumption (Visit 4) | -7.74 (12.87) | 1.59 (12.38)
  Prospective food consumption (Visit 5): number analyzed (Participants) | 28 | 26
  Prospective food consumption (Visit 5) | -6.18 (16.92) | 4.23 (14.46)
  Hunger (Visit 4): number analyzed (Participants) | 28 | 26
  Hunger (Visit 4) | -3.71 (7.97) | 2.13 (10.88)
  Hunger (Visit 5): number analyzed (Participants) | 28 | 26
  Hunger (Visit 5) | -3.41 (8.96) | 2.63 (13.00)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Satiety (Visit 4); Test type: Superiority; p = 0.1768, Mixed Models Analysis; Least Square Mean Difference = 3.98, 95% CI 2-sided [-1.85 to 9.82], Standard Error of Mean 2.91
Statistical Analysis 2: Comparison: Liraglutide vs Placebo; Satiety (Visit 5); Test type: Superiority; p = 0.1137, Mixed Models Analysis; Least Square Mean Difference = 3.43, 95% CI 2-sided [-0.85 to 7.70], Standard Error of Mean 2.13
Statistical Analysis 3: Comparison: Liraglutide vs Placebo; Fullness (Visit 4); Test type: Superiority; p = 0.1858, Mixed Models Analysis; Least Square Mean Difference = 2.85, 95% CI 2-sided [-1.41 to 7.11], Standard Error of Mean 2.12
Statistical Analysis 4: Comparison: Liraglutide vs Placebo; Fullness (Visit 5); Test type: Superiority; p = 0.5288, Mixed Models Analysis; Least Square Mean Difference = 1.41, 95% CI 2-sided [-3.05 to 5.86], Standard Error of Mean 2.22
Statistical Analysis 5: Comparison: Liraglutide vs Placebo; Prospective food consumption (Visit 4); Test type: Superiority; p = 0.0054, Mixed Models Analysis; Least Square Mean Difference = -8.46, 95% CI 2-sided [-14.30 to -2.61], Standard Error of Mean 2.91
Statistical Analysis 6: Comparison: Liraglutide vs Placebo; Prospective food consumption (Visit 5); Test type: Superiority; p = 0.0117, Mixed Models Analysis; Least Square Mean Difference = -9.78, 95% CI 2-sided [-17.29 to -2.27], Standard Error of Mean 3.75
Statistical Analysis 7: Comparison: Liraglutide vs Placebo; Hunger (Visit 4); Test type: Superiority; p = 0.0093, Mixed Models Analysis; Least Square Mean Difference = -6.58, 95% CI 2-sided [-11.48 to -1.69], Standard Error of Mean 2.44
Statistical Analysis 8: Comparison: Liraglutide vs Placebo; Hunger (Visit 5); Test type: Superiority; p = 0.0296, Mixed Models Analysis; Least Square Mean Difference = -6.39, 95% CI 2-sided [-12.12 to -0.66], Standard Error of Mean 2.86

9. Secondary Outcome: Change From Baseline in Area Under the Plasma Concentration-Time Profile of Acetaminophen for 0-60 Minutes and 0-300 Minutes (AUC0-60min and AUC0-300min) After Acetaminophen Dose at Visits 4 and 5
Description: A non investigational medicinal product (acetaminophen 1.5 gram [g]) was administered as a challenge agent for the assessment of gastric emptying. The blood sampling for determining acetaminophen concentrations was performed at 7 time points: prior to breakfast and at 30, 60, 90, 120, 180 and 300 minutes after intake of the acetaminophen with breakfast. Baseline was calculated at Visit 3 (Study Day -1).
Time Frame: Prior to breakfast and at 30,60,90,120,180 and 300 minutes after intake of the acetaminophen with breakfast on Visit 3,Visit 4 (Study Day 20) and Visit 5 (Study Day 41)
Population: Number of participants analyzed includes participants who met the criteria: completed baseline assessment of food intake;received at least 1 dose of randomized, blinded IP;completed at least 1 post baseline measurement(after taking randomized IP).Number analyzed includes participants contributing to AUC0-60min and AUC0-300min at specified visits.
Measure: Mean (Standard Deviation); unit: microgram*minute/milliliter (ug*min/mL)
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 30 | 26
microgram*minute/milliliter (ug*min/mL)
  AUC0-60min (Visit 4) | 18.30 (204.93) | -4.55 (262.11)
  AUC0-60min (Visit 5): number analyzed (Participants) | 28 | 26
  AUC0-60min (Visit 5) | 81.19 (166.47) | -8.28 (258.55)
  AUC0-300min (Visit 4): number analyzed (Participants) | 29 | 26
  AUC0-300min (Visit 4) | 197.79 (491.11) | -12.92 (489.50)
  AUC0-300min (Visit 5): number analyzed (Participants) | 27 | 26
  AUC0-300min (Visit 5) | 394.22 (401.62) | 47.31 (564.52)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; AUC0-60min (Visit 4); Test type: Superiority; p = 0.5008, Mixed Models Analysis; Least Square Mean Difference = 35.56, 95% CI 2-sided [-69.64 to 140.76], Standard Error of Mean 52.46
Statistical Analysis 2: Comparison: Liraglutide vs Placebo; AUC0-60min (Visit 5); Test type: Superiority; p = 0.0348, Mixed Models Analysis; Least Square Mean Difference = 106.15, 95% CI 2-sided [7.86 to 204.44], Standard Error of Mean 48.95
Statistical Analysis 3: Comparison: Liraglutide vs Placebo; AUC0-300min (Visit 4); Test type: Superiority; p = 0.1040, Mixed Models Analysis; Least Square Mean Difference = 214.24, 95% CI 2-sided [-45.59 to 474.07], Standard Error of Mean 129.48
Statistical Analysis 4: Comparison: Liraglutide vs Placebo; AUC0-300min (Visit 5); Test type: Superiority; p = 0.0152, Mixed Models Analysis; Least Square Mean Difference = 348.43, 95% CI 2-sided [70.20 to 626.66], Standard Error of Mean 138.29

ADVERSE EVENTS:
Time Frame: From Baseline (Visit 3, Study Day -1 and Day 0) to Day 73.
Description: The same event may appear as both an AE and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonseriousevent during the study.
Arm/Group | Liraglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/28
Other Adverse Events (participants affected / at risk) | 30/32 | 18/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Liraglutide (N=32) | Placebo (N=28)
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 6 | 1
Constipation (Gastrointestinal disorders) | 9 | 3
Diarrhoea (Gastrointestinal disorders) | 11 | 4
Dyspepsia (Gastrointestinal disorders) | 7 | 2
Nausea (Gastrointestinal disorders) | 15 | 1
Vomiting (Gastrointestinal disorders) | 6 | 0
Injection site bruising (General disorders) | 7 | 4
Injection site erythema (General disorders) | 4 | 0
Injection site mass (General disorders) | 2 | 0
Injection site pain (General disorders) | 2 | 0
Injection site pruritus (General disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 8 | 2
Headache (Nervous system disorders) | 11 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0
Eructation (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dizziness (Nervous system disorders) | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Amylase increased (Investigations) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 4
Urinary tract infection (Infections and infestations) | 2 | 0
Asthenia (General disorders) | 2 | 0
Fatigue (General disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-11-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT03041792/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-16): https://cdn.clinicaltrials.gov/large-docs/92/NCT03041792/SAP_001.pdf